CLINICAL TRIAL: NCT00672412
Title: A Phase I/II Comparative Pharmacokinetic Study of the Fixed-Dose Combination (FDC) of Zidovudine (ZDV), Lamivudine (3TC), and Nevirapine (NVP) as GPO-Vir Z30 Pediatric Tablets Versus the Individual Liquid Formulations in HIV-Infected Children Greater Than or Equal to Five Months and Less Than 13 Years of Age in Thailand
Brief Title: Safety and Pharmacokinetic Study of Fixed Dose Combination of Zidovudine, Lamivudine, and Nevirapine in HIV-Infected Children in Thailand
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P1069; 10620 (Registry Identifier: DAIDS ES); IMPAACT P1069
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2012-09

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Lamivudine; Nevirapine; Zidovudine

ARMS (2):
- 1 (Experimental): Participants receive GPO-VIR Z30 tablets containing ZDV, 3TC, and NVP for the first 14 days of the study. On Day 15, participants receive liquid ZDV, 3TC, and NVP for the following 14 days of the study.
  Interventions: Drug: GPO-Vir Z30 tablet; Drug: Lamivudine; Drug: Nevirapine; Drug: Zidovudine
- 2 (Experimental): Participants receive liquid ZDV, 3TC, and NVP for the first 14 days of the study. On Day 15, participants receive GPO-VIR Z30 tablets containing ZDV, 3TC, and NVP for the following 14 days of the study.
  Interventions: Drug: GPO-Vir Z30 tablet; Drug: Lamivudine; Drug: Nevirapine; Drug: Zidovudine

INTERVENTIONS:
Drug: GPO-Vir Z30 tablet — Tablet consisting of ZDV 30 mg/3TC 15 mg/NVP 28 mg taken orally twice daily
Drug: Lamivudine — Oral suspension containing 10 mg 3TC in each mL. Dosage depends on weight.
  Other Names: 3TC; Epivir
Drug: Nevirapine — Oral solution containing 10 mg NVP in each mL. Dosage depends on weight.
  Other Names: NVP; Viramune
Drug: Zidovudine — Oral solution containing 10 mg ZDV in each mL. Dosage depends on weight.
  Other Names: ZDV; Retrovir

SUMMARY:
In 2005, there were 50,620 HIV-infected children living in Thailand. Current anti-HIV regimens, comprised of individual pills for each drug, frequently lead to missed doses. To properly control their infection, regimens that are tolerable and effective in children and without pill burden are necessary. The primary purpose of this study is to evaluate the safety and bioavailability of GPO-VIR Z30, a combination fixed dose tablet containing zidovudine (ZDV), lamivudine (3TC), and nevirapine (NVP), in HIV-infected children in Thailand.

DETAILED DESCRIPTION:
An important factor affecting the therapeutic response to ARVs is adherence. A common reason for poor adherence is high pill burden. A combination fixed dose drug approach appears to be an effective strategy to improve adherence and therapeutic response. In this study, investigators will compare the bioavailability and safety of GPO-VIR Z30, a combination fixed dose drug, with the liquid formulations of ZDV,3TC, and NVP, in children.

This study will last approximately 8 weeks. Participants will be randomly assigned to one of two arms. Participants in Arm 1 will receive GPO-VIR Z30 for 2 weeks before receiving liquid formulations of ZDV, 3TC, and NVP for the following 2 weeks. Participants in Arm 2 will receive liquid formulations of ZDV, 3TC, and NVP for 2 weeks before receiving GPO-VIR Z30 for the following 2 weeks.

This study will consist of 4 study visits after screening. Visits will occur at study entry and on Days 14, 28, and 56. Medical history and a physical exam will occur at all visits. A pregnancy test will occur for females at all visits. Pharmacokinetic tests, involving hospitalization for the 12 hour procedure, will occur on Days 14 and 28. Safety and adherence monitoring will occur by telephone on Days 7, 11 or 12, 13, 21, 25 or 26, 27, and 35. Home visits for directly observed therapy (DOT) may also occur.

ELIGIBILITY:
Inclusion Criteria:

* Weigh between 6 and 30 kilograms
* HIV infected
* Receiving HAART regimen of NVP and 2 NRTIs. More information on this criterion can be found in the protocol.
* Agree to use two appropriate forms of contraception. More information on this criterion can be found in the protocol.
* Ability to swallow study drugs
* Willing to be hospitalized for 12-hour intensive PK study
* Agree to use two appropriate forms of contraception. More information on this criterion can be found in the protocol.
* Parent or legal guardian able and willing to provide written informed consent

Exclusion Criteria:

* Certain abnormal laboratory values. More information on this criterion can be found in the protocol.
* Vomiting or diarrhea (greater than Grade 2) within 30 days prior to study entry
* History of immunologic failure. More information on this criterion can be found in the protocol.
* Current treatment for an acute serious bacterial, viral, or opportunistic infection
* History of dose-limiting toxicity requiring treatment discontinuation of any of the study drugs
* Hypersensitivity to study drugs
* Surgical or medical problem affecting gastrointestinal motility or absorption or liver function
* Treatment with experimental drugs within 30 days prior to study entry
* Acute hepatitis
* Chemotherapy for active malignancy
* Any clinically significant diseases or findings during the screening medical history or physical examination that, in the opinion of the investigator, may interfere with the study
* Pregnant

Ages: 5 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety and comparative bioavailability measured by concentration difference between the GPO-Vir Z30 and standard liquid regimens | Throughout study
Therapeutic adequacy of NVP measured by treatment-specific concentration distributions | Throughout study

SECONDARY OUTCOMES:
Comparisons in PK analyses between GPO-VIR Z30 and standard liquid regimens including pharmacokinetic parameters, adverse drug reactions, and the influence of SNPs on NVP pharmacokinetic parameters | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Kulkanya Chokephaibulkit, MD, Study Chair — Siriraj Hospital; Nirum Vanprapar, MD, Study Chair — Siriraj Hospital; Ram Yogev, MD, Study Chair — CMRC Children's Memorial Hospital
Locations (4):
- Thailand (4):
  - Prapokklao Hosp. CRS, Muang District, Changwat Chanthaburi
  - Siriraj Hospital Mahidol University CRS, Bangkok, Ratchathewi
  - Chiang Mai University Pediatrics-Obstetrics CRS, Chiang Mai
  - Chonburi Hosp. CRS, Chon Buri

REFERENCES:
- [Background] Kiertiburanakul S, Khongnorasat S, Rattanasiri S, Sungkanuparph S. Efficacy of a generic fixed-dose combination of stavudine, lamivudine and nevirapine (GPO-VIR) in Thai HIV-infected patients. J Med Assoc Thai. 2007 Feb;90(2):237-43. PMID 17375626
- [Background] Manosuthi W, Kiertiburanakul S, Chaovavanich A, Sungkanuparph S. Plasma nevirapine levels and 24-week efficacy of a fixed-dose combination of stavudine, lamivudine and nevirapine (GPO-VIR) among Thai HIV-infected patients. J Med Assoc Thai. 2007 Feb;90(2):244-50. PMID 17375627